CLINICAL TRIAL: NCT03439995
Title: Goal of Open Lung Ventilation in Donors
Acronym: GOLD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial no longer feasible
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of California, San Francisco (Other); University of California, Los Angeles (Other); Stanford University (Other); Donor Network West (Unknown)
Responsible Party: Principal Investigator, Lorraine B. Ware, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL126176 (NIH)
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Brain Death; Organ Donation; Organ Transplant Failure or Rejection
MeSH Terms: conditions — Brain Death; Rejection, Psychology

STUDY DESIGN:
Intervention Model Description: Enrolled donors will be randomly assigned to two different modes of mechanical ventilation for the duration of donor management
Who Masked: Outcomes Assessor
Masking Description: Outcomes in donors and lung transplant recipients will be done by assessors who are blinded to ventilator treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Lung Protective Ventilation (Experimental): Volume cycled assist control ventilation with tidal volume 8 cc/kg predicted body weight, PEEP 10 cm water (H2O), recruitment maneuvers every 8 hours and after any ventilator disconnect
  Interventions: Other: Open lung protective ventilation
- Conventional Ventilation (Active Comparator): Volume cycled assist control ventilation with tidal volume 10 cc/kg predicted body weight, PEEP 5 cm H2O, recruitment maneuvers after any ventilator disconnect
  Interventions: Other: Conventional ventilation

INTERVENTIONS:
Other: Open lung protective ventilation — Higher PEEP, lower tidal volume mechanical ventilation
  Arms: Open Lung Protective Ventilation
Other: Conventional ventilation — Lower PEEP, standard tidal volume mechanical ventilation
  Arms: Conventional Ventilation

SUMMARY:
The primary goal of this study is to assess whether ventilation of deceased organ donors with an open lung protective ventilatory strategy will improve donor lung utilization rates and donor oxygenation compared to a conventional ventilatory strategy.

DETAILED DESCRIPTION:
Deceased organ donors are maintained on life support including mechanical ventilation during the time between brain death and organ procurement. The optimal mode of mechanical ventilation for deceased organ donors has not been definitively established. Since deceased organ donors may develop atelectasis leading to impaired oxygenation, an open lung protective ventilatory strategy with higher positive end expiratory pressure (PEEP), lower tidal volume and recruitment maneuvers has been hypothesized to be beneficial. Favorable outcomes were observed in a European clinical trial comparing open lung protective ventilation (OLPV) to a conventional ventilatory strategy in terms of donor oxygenation and lung utilization for transplantation (Mascia L et al, Journal of the American Medical Association 2010). However, donor management procedures in Europe are much shorter in duration compared to the US and it is not clear that these findings are generalizable to the US donor management environment.

The GOLD trial will test the effect of an OLPV strategy compared to conventional ventilation (CV) in the US donor management environment. This multi center trial will enroll 400 brain dead organ donors randomized into 1 of 2 treatment arms. After randomization, mechanical ventilation will be protocolized according to treatment arm with one arm receiving control ventilation (CV) utilizing standard Donor Network West (DNW) protocols and the other arm receiving the OLPV strategy with higher positive end expiratory pressure (PEEP) and lower tidal volume compared to CV. The primary outcomes is donor lung utilization for transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Brain death
* Authorization for research
* ≥13 years of age

Exclusion Criteria:

* Arterial/Inspired oxygen ratio (PaO2/FiO2) ≤ 150 mmHg
* PaO2/FiO2 ≥ 400 mmHg
* BMI > 40
* Hepatitis B surface antigen positive
* Hepatitis C positive
* Failure to complete donation process
* Hemodynamic instability

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Donor lung utilization rate | during donor management period (usually 12-48 hours)
  Percent of donor lungs procured and transplanted into recipient

SECONDARY OUTCOMES:
Donor lung utilization in likely donors | during donor management period (usually 12-48 hours)
  Percent of donor lungs used from donors with < 50 pack year smoking, age < 65, negative serologies, and no underlying chronic lung disease
Donor oxygenation | during donor management period (usually 12-48 hours)
  Change in donor arterial oxygen (PaO2) from enrollment to procurement
Donor static compliance of the respiratory system | during donor management period (usually 12-48 hours)
  Change in compliance of the respiratory system (in ml/cm H2O) from enrollment to procurement. Static compliance (Cstat) is calculated as Cstat = ΔV / Pplat - PEEP where V is the volume delivered by the ventilator, Pplat is the end-inspiratory plateau pressure and PEEP is the level of positive end expiratory pressure.
Donor radiographic atelectasis scoring | during donor management period (usually 12-48 hours)
  Change in chest radiograph atelectasis score from enrollment to procurement
Recipient primary graft dysfunction | 72 hours after transplant
  International Society of Heart and Lung Transplantation grade 2 or 3 primary graft dysfunction in lung transplant recipient
Recipient mortality | 30 days after transplant
  Lung transplant recipient death

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine B Ware, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (4):
- United States (4):
  - UCLA, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Donor Network West, San Ramon, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mascia L, Pasero D, Slutsky AS, Arguis MJ, Berardino M, Grasso S, Munari M, Boifava S, Cornara G, Della Corte F, Vivaldi N, Malacarne P, Del Gaudio P, Livigni S, Zavala E, Filippini C, Martin EL, Donadio PP, Mastromauro I, Ranieri VM. Effect of a lung protective strategy for organ donors on eligibility and availability of lungs for transplantation: a randomized controlled trial. JAMA. 2010 Dec 15;304(23):2620-7. doi: 10.1001/jama.2010.1796. PMID 21156950
- [Derived] Ware LB, Koyama T, Shaver CM, Swain S, Nguyen J, Salehi A, Dhillon G, Wickersham N, Maheshwari J, Singer JP, Weigt SS, Kukreja J, Matthay MA. A randomized trial of open lung protective ventilation compared to conventional mechanical ventilation in deceased organ donors. J Heart Lung Transplant. 2025 Aug;44(8):1251-1259. doi: 10.1016/j.healun.2025.03.027. Epub 2025 Apr 3. PMID 40187505